CLINICAL TRIAL: NCT01343420
Title: Dog Hair Evaluation Potency by Prick Skin Testing
Brief Title: Dog Hair Extract Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Jewish Health (Other)
Collaborators: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: ALK-Abelló Dog Allergen
Record Dates: First submitted 2011-04-26; First posted 2011-04-28 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Potency of Dog Hair Extract
Keywords: Skin tests; Dog Hair; Allergy Extract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dog Hair Extract, ALK-Abelló, Inc. (Active Comparator)
  Interventions: Biological: Dog Hair Extract, ALK-Abelló, Inc.

INTERVENTIONS:
Biological: Dog Hair Extract, ALK-Abelló, Inc. — ALK-Abelló dog epithelial 1:10w/v glycerin

SUMMARY:
Liquid allergen extracts contain proteins, such as (but not limited to) tree, weed, cat, cockroach, and nuts, and are used to identify allergies by observing the body's reaction to the introduction of extract underneath the skin. There are a few dog allergen extracts commercially available in the US for allergy testing; however, none of these products are standardized, meaning they are not required to be the same strength. Because some extracts are not as potent (strong) as others, it's possible that some patients' allergies are misdiagnosed. Typically, the most potent (strong), but safe extract should be used so that allergic patients are correctly diagnosed.

The purpose of this study is to compare the safety and potency of an investigational (not approved for use by the United States Food and Drug Administration [FDA]) dog allergen extract with two commercially available dog extracts, which are of differing potencies.

DETAILED DESCRIPTION:
This study is designed to assess the potency of a modified dog hair and dander extract in comparison with the two commercially available dog hair and dander extracts. This is a pilot study to estimate a target strength of dog extract in order to proceed to further studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients must sign informed consent before completing any study procedure.
* Age 18 years and ≤60 years.
* Dog-sensitized patients as indicated by a mean wheal > 5 mm with the AP dog extract.
* Females of child-bearing potential must have a negative pregnancy test the day of skin testing.
* Patients who are able to understand the information given and be compliant with the protocol.

Exclusion Criteria:

* Asthma requiring treatment with medications other than beta-2 inhaled agonists and montelukast inhibitors.
* Patients with a history of asthma or wheezing with an FEV1 <80%.
* Subjects who have taken an ocular or nasal antihistamine within 5 days prior to the procedures.
* Patients who have received any desensitization for dog allergen in the past 5 years.
* Patients with any past or current clinically significant condition that may affect the patient's participation or the outcome of the study to the discretion of the investigator. These include, but are not limited to, anaphylaxis with cardio-respiratory symptoms, chronic urticaria and angioedema unless related to dog exposure, severe atopic dermatitis, malignancy, cardiovascular, hepatic, renal, hematological, neurological, immunological, and endocrine disease.
* Subjects taking beta blockers, ace inhibitors, continuous systemic corticotherapy, immunosuppressive drugs or monoamine oxidase inhibitors.
* Use of H1 antagonists, tricyclic antidepressants and phenothiazines within 5 days prior to the testing.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2010-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
End-point dilution giving a positive prick skin test in dog allergic subjects. | Study Completion
  The concentration of each allergen extract which produced a 5 mm wheal for each subject will be calculated. From this, the relative potency of each extract will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Harold Nelson, M.D., Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States